CLINICAL TRIAL: NCT05990361
Title: Comparison of Sexual Function, Body Image, Kinesiophobia and Physical Activity Level in Women With and Without Pregnancy-related Pelvic Girdle Pain''
Brief Title: Sexual Function, Body Image, Kinesiophobia and Physical Activity in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Other Study IDs: 18.04.2023-90204
Record Dates: First submitted 2023-05-09; First posted 2023-08-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy-Related Pelvic Girdle Pain
Keywords: pelvic girdle pain; sexual function; body image; fear of movement
MeSH Terms: conditions — Pelvic Girdle Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with pelvic girdle pain: The subjects who have at least one positive result from Active Straight Leg Raise, and Posterior Pelvic Pain Provocation Tests; and at least two positive results from the Pelvic Compression and Distraction, Patrick Faber, Gaenslen and Long Dorsal Sacroiliac Ligament Palpation tests are classified as with PGP group.
  Interventions: Diagnostic Test: clinical diagnostic test
- women without pelvic girdle pain: The subjects who have not at least one positive result from Active Straight Leg Raise, and Posterior Pelvic Pain Provocation Tests; and at least two positive results from the Pelvic Compression and Distraction, Patrick Faber, Gaenslen and Long Dorsal Sacroiliac Ligament Palpation tests are classified as without PGP group.
  Interventions: Diagnostic Test: clinical diagnostic test

INTERVENTIONS:
Diagnostic Test: clinical diagnostic test — The clinical diagnosis tests are Active Straight Leg Rise ASLR, Posterior Pelvic Pain Provocation, Long Dorsal Sacroiliac Ligament Palpation (LDSLP), Pelvic Compression, Pelvic Distraction, Patrick-Faber Test (PF), and Gaenslen Test (GT).
  The subjects who had at least one positive result from ASLR and P4 Tests; and at least two positive results from the Pelvic Compression and Distraction, PF, GT and LDSLP tests are classified as with PGP group.

SUMMARY:
This study compares sexual function, body image, kinesiophobia and physical activity level in women with and without pregnancy-related pelvic girdle pain.

DETAILED DESCRIPTION:
Pelvic girdle pain (PGP) is a condition felt around the posterior iliac crystals, gluteal region and the sacroiliac joints, may spread to the back of the thigh, and may occur together or separately with pain in the symphysis pubis. Pregnancy-related PGP causes problems in the sexual life of women. Body image differs with the development of physical symptoms and changes in body size and shape during pregnancy. Body dissatisfaction resulting from physical changes can cause problems in women's attitudes towards sexuality. Sexual function is affected by physiological, anatomical and psychological changes that occur during pregnancy. Sexual function during pregnancy has been associated with conditions such as body image, physical activity level, and pain.

In the literature, there are studies evaluating the relationship between sexual function and body image in pregnant women and in different populations. However, in these studies, questionnaires specific to pregnant women were not used to evaluate sexual function and body image, and a comparison of these parameters was not investigate in women with and without pregnancy-related PGP.

Therefore, this study was planned to compare sexual function, body image, kinesiophobia and physical activity levels in women with and without pregnancy-related PGP.

The outcome measures are Pregnancy Sexual Response Inventory (PSRI), Body Image in Pregnancy Scale (BIPS-Turkish), Tampa Kinesiophobia Scale (TKS) and Pregnancy physical activity questionnaire (PPAQ).

The clinical diagnosis tests are Active Straight Leg Rise, Posterior Pelvic Pain Provocation Test, Long Dorsal Sacroiliac Ligament Palpation, Pelvic Compression, Pelvic Distraction, Patrick-Faber Test and Gaenslen Test.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 40 years-old,
* Being second or third trimester of pregnancy
* Being literate in Turkish

Exclusion Criteria:

* Having a pregnancy complication (preeclampsia, pregnancy-induced hypertension, diabetes, etc.),
* Having a known gynecological or urological problem that may mimic PGP
* Having neurological (multiple sclerosis, spinal cord injury, etc.), orthopedic (hip dislocation, etc.), cardiopulmonary (heart failure, chronic obstructive pulmonary disease, etc.) problems that affect sexual function and physical activity,
* Having situations in which sexual activity is contraindicated and should be restricted (placenta previa, risk of premature birth, cervical insufficiency, antepartum hemorrhage, premature rupture of membranes, genital infection, etc.),
* Having visual, auditory and cognitive problems that may prevent participation in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with and without pregnancy-related pelvic girdle pain
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy Sexual Response Inventory-Turkish version | immediately before the clinical diagnostic tests will be applied the questionnaire
  to assess sexual functions in pregnant women with and without PGP
Body Image in Pregnancy Scale (BIPS-Turkish) | immediately before the clinical diagnostic tests will be applied the questionnaire
  to evaluate body image perceptions of Turkish pregnant women with and without PGP
Tampa Scale for Kinesiophobia-Turkish version | immediately before the clinical diagnostic tests will be applied the questionnaire
  to evaluate level of kinesiophobia of Turkish pregnant women with and without PGP
Pregnancy Physical Activity Questionnaire-Turkish version | immediately before the clinical diagnostic tests will be applied the questionnaire
  To evaluate the physical activity level of pregnant women with and without PGP

SECONDARY OUTCOMES:
Pelvic Girdle Questionnaire Pelvic Girdle Questionnaire-Turkish version | immediately after the clinical diagnostic tests for PGP will be applied the questionnaire
  To evaluate both disability and symptoms women with pregnancy-related PGP

CONTACTS AND LOCATIONS:
Overall Officials: SEMİHA YENİŞEHİR, Principal Investigator — Muş Alparslan University
Locations (1):
- Semiha Yenişehir, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yenisehir S, Karakaya IC, Ozbey G. Sexual Function of Women with and without Pregnancy-Related Pelvic Girdle Pain and its Relationship with Physical Activity, Kinesiophobia and Body Image: A Cross-Sectional Comparative Study. Reprod Sci. 2024 Oct;31(10):3122-3131. doi: 10.1007/s43032-024-01644-2. Epub 2024 Jul 9. PMID 38981994